CLINICAL TRIAL: NCT02450734
Title: Safety and Efficiency of Ultrasound-guided Intermediate Cervical Plexus Block for Carotid Surgery
Brief Title: Ultrasound-guided Intermediate Cervical Plexus Block for Carotid Surgery
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: IMM CEPAR : 2012-014
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Carotid Artery Stenosis
Keywords: ultrasound-guided intermediate cervical plexus block
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: Realisation of an ultrasound-guided intermediate cervical plexus block for anesthesia of carotid endarterectomy
  Interventions: Procedure: Ultrasound-guided intermediate cervical plexus block

INTERVENTIONS:
Procedure: Ultrasound-guided intermediate cervical plexus block

SUMMARY:
Since stroke and myocardial ischemia are major causes of perioperative morbidity and mortality associated with carotid endarterectomy, monitoring the brain and ensuring the best hemodynamic stability are important goals of perioperative management.

The investigators conducted a prospective observational study about efficacy and safety of the ultrasound-guided intermediate cervical plexus block (CPB), with early (immediate postoperative) and mid-term (day 30) outcomes in awake patients undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
From April 2011 to May 2013, all patients undergoing a carotid endarterectomy were informed of the study and prospectively included. The study was approved by our institutional ethical Review Board (CEPAR, Institut Mutualiste Montsouris Paris France). Oral consent was obtained from patients. Written informed consent of the patients to participate was not necessary according to the French law regarding observational study.

The anesthesiologist in charge of the patient recorded all the parameters of the ultrasound-guided intermediate cervical plexus block: facility and duration of block performance, local anesthetic volume, quality of anesthesia and surgical dissection, and adverse effects of the intermediate CPB. . Neurological status was assessed intraoperatively, in the postoperative setting and at one month after the procedure. Perioperative hemodynamic stability (intraoperative non invasive blood pressure variations) and pulse oxymetry were recorded. As well as ECG and cardiac Troponin I (cTnI) measurments performed the day before surgery and each morning during the 3 first postoperative days. Any clinical coronary or neurological event was recorded at one month.

Statistical analysis was performed on Prism 6 for Mac OS X (Version 6.0c, www.graphpad.com). Data are presented as mean ± standard deviation (SD) for continuous data and number (percentage) for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
quality of anesthesia | immediate
  assessed by the patient (quality scale) and absence of the need to general anesthesia

SECONDARY OUTCOMES:
Hemodynamic stability | immediate during surgery
  measurements of non invasive arterial pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LEBLANC, Doctor, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Department of Anesthesia Institut Mutualiste Montsouris, Paris, Paris, France

REFERENCES:
- [Result] Schechter MA, Shortell CK, Scarborough JE. Regional versus general anesthesia for carotid endarterectomy: the American College of Surgeons National Surgical Quality Improvement Program perspective. Surgery. 2012 Sep;152(3):309-14. doi: 10.1016/j.surg.2012.05.008. Epub 2012 Jun 27. PMID 22749369
- [Result] Usui Y, Kobayashi T, Kakinuma H, Watanabe K, Kitajima T, Matsuno K. An anatomical basis for blocking of the deep cervical plexus and cervical sympathetic tract using an ultrasound-guided technique. Anesth Analg. 2010 Mar 1;110(3):964-8. doi: 10.1213/ANE.0b013e3181c91ea0. Epub 2009 Dec 15. PMID 20008914
- [Result] Choquet O, Dadure C, Capdevila X. Ultrasound-guided deep or intermediate cervical plexus block: the target should be the posterior cervical space. Anesth Analg. 2010 Dec;111(6):1563-4; author reply 1564-5. doi: 10.1213/ANE.0b013e3181f1d48f. No abstract available. PMID 21106978